CLINICAL TRIAL: NCT03344159
Title: Spironolactone Therapy in Chronic Stable Right HF Trial
Acronym: STAR-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170694
Record Dates: First submitted 2017-09-28; First posted 2017-11-17 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Chronic Right-Sided Heart Failure; Pulmonary Arterial Hypertension; Pulmonary Hypertension, Primary, 2; Pulmonary Hypertension, Primary, 3; Pulmonary Hypertension, Primary, 4; Cardiomyopathy Right Ventricular
Keywords: Mineralocorticoid receptor antagonist; Brain natriuretic peptide (BNP); Sympathetic Nervous System; Positron Emissions Tomography
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Lipodystrophy, Congenital Generalized, Type 3 | interventions — Spironolactone; Rubidium-82

STUDY DESIGN:
Intervention Model Description: STAR-HF is a phase 4 single center, randomized, placebo controlled trial comparing spironolactone 12.5mg daily up to a maximum dose of 50 mg daily if tolerated to matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be blinded to study treatment for the duration of the study. Clinicians will also be blinded to study drug assignment. Evaluation of all study results will be done blinded to treatment randomization. Because of the double-blind design, safety laboratory tests, and monitoring of potential side effects will be performed for each participant for the duration of the trial, regardless of the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spironolactone (Experimental): Participants with chronic right-sided heart failure will receive spironolactone 12.5mg daily up to a maximum dose of 50 mg daily for a total duration of 12 weeks.
  Interventions: Drug: Spironolactone; Radiation: PET/CT Scan: Two PET scans using 1. C-11 HED and 2. N-13 Ammonia or rubidium-82; Diagnostic Test: Cardiac MRI (Gadolinium enhanced)
- Placebo (Placebo Comparator): Participants with chronic right-sided heart failure will receive placebo daily for a total duration of 12 weeks.
  Interventions: Drug: Placebo; Radiation: PET/CT Scan: Two PET scans using 1. C-11 HED and 2. N-13 Ammonia or rubidium-82; Diagnostic Test: Cardiac MRI (Gadolinium enhanced)

INTERVENTIONS:
Drug: Spironolactone — Spironolactone 12.5mg daily up to a maximum dose of 50 mg daily if tolerated for a total duration of 12 weeks.
  Arms: Spironolactone
Drug: Placebo — Placebo daily for a total of duration of 12 weeks
  Arms: Placebo
Radiation: PET/CT Scan: Two PET scans using 1. C-11 HED and 2. N-13 Ammonia or rubidium-82 — At baseline and 12 weeks, all participants will undergo rest perfusion PET imaging according to standard protocols with either 82-Rb or N-13 NH3, followed by C-11 HED PET.
Diagnostic Test: Cardiac MRI (Gadolinium enhanced) — At baseline and 12 weeks all participants will undergo cMR to assess RV function and structure. We will acquire precontrast T2 and native T1 maps, and post gadolinium T1 maps.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and mechanistic effects of spironolactone, an aldosterone receptor antagonist, on sympathetic nervous system activity and right heart function and remodeling in patients with chronic right heart failure.

DETAILED DESCRIPTION:
This study is a phase 4, single center, randomized, double blind, placebo-controlled trial evaluating the safety, tolerability and mechanistic effects of spironolactone, an aldosterone antagonist, on neurohormonal activity and remodeling in patients with chronic right heart failure (RHF).

RHF is one of the most important predictors of prognosis in many cardiac disease states including pulmonary hypertension (PH), and left heart failure. Sympathetic nervous system activation plays an important role in the development and progression of heart failure. It remains to be determined whether there is a role for neurohormonal therapy in chronic right HF, but evidence points to the role of sympathetic nervous system stimulation and activation of the renin-angiotensin and aldosterone system as a contributor to progressive right heart failure.

The study will determine if treatment with spironolactone is associated with reduction in right ventricular wall stress. In addition, the study aims to evaluate the effects of spironolactone on cardiac sympathetic activity assessed by HED(11 C-hydroxy-ephedrine) retention on PET(positron emission tomography) imaging, and global autonomic function assessed by heart rate variability.

Approximately 30 patients with RHF will be randomized to receive either spironolactone daily or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provide a personally signed and dated inform consent form.
* Male or female ≥ 18 years.
* Able to comply with all study procedures.
* History of right heart failure (RHF) secondary to either:

  i) WHO, group 1 pulmonary arterial hypertension PAH OR ii) WHO group II PH with normal LV systolic function OR iii) WHO group III or IV PH OR iv) primary RV cardiomyopathy.
* Current NYHA II-IV
* RV dysfunction as measured by 2D echocardiogram:

  i)defined as a tricuspid annular plane systolic excursion (TAPSE) <16 mm ii) and /or a two dimensional fractional area change <35% on screening echo plus
* NT-proBNP>400 pg/ml
* Chronic use of diuretics
* Clinical stability: defined as no need for increased diuretics, hospitalization or emergency room visit 3 months prior to enrollment

Exclusion Criteria:

* Patients on chronic MRA therapy or other potassium sparing diuretics.
* Baseline serum potassium>5 ummol/l.
* Estimated glomerular filtration rate <30 ml/min.
* LV ejection fraction <45%,
* Moderate or severe LV diastolic function,
* Moderate or severe aortic or valvular disease.
* Patients requiring augmentation of diuretics or otherwise not meeting definition for clinical stability.
* Severe Liver Failure (Child-Pugh Class C)
* Claustrophobia or inability lie still in a supine position
* Patients with contraindications to either PET or CMR imaging
* Pregnancy or lactation.
* Unable to provide consent and comply with follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Ventricular Wall Stress | Baseline and 12 weeks
  To determine if treatment with spironolactone is associated with a significant reduction in RV ventricular wall stress, as reflected by a reduction in serum NT-proBNP, in patients with chronic stable right HF when compared to placebo.

SECONDARY OUTCOMES:
Change in Cardiac Sympathetic Nervous System Activity | Baseline to 12 weeks
  Changes in cardiac sympathetic activity, as assessed by an increase in 11[C]-hydroxy-ephedrine (HED) retention by cardiac PET imaging.
Change in Cardiac Autonomic Nervous System Function | Baseline to 12 weeks
  Heart rate variability
Change in Systemic Sympathetic Activation | Baseline to 12 weeks
  Changes in plasma levels of epinephrine and norepinephrine
Change in Right Ventricle Structure | Baseline to 12 weeks
  Changes in RV end-diastolic and end-systolic size.
Change in Right Ventricle Function | Baseline to 12 weeks
  Changes in RV ejection fraction
Change in Right Ventricle areas of fibrosis | Baseline to 12 weeks
  Changes in RV areas of fibrosis assessed with T1 weighted MR imaging.
Number of participants with treatment-related adverse events. | number of adverse events from baseline to 12 weeks.
  1. incidence of worsening renal function (defined as a change in estimated glomerular filtration rate>30%). 2. Incidence of hyperkalemia (>4.5, 5 or 5.5 mmol/L)
Change in Biomarkers of Fibrosis | Baseline to 12 weeks
  Changes in biomarkers of fibrosis (ST2, PIINP, CITB, TIMP1, MMP-9)

OTHER OUTCOMES:
Change in Serum Aldosterone | Baseline to 12 weeks
  changes in plasma levels of aldosterone
Change in Six Minute walk test | Baseline, 6 weeks, 12 weeks
  Distance a participant can walk in a period of 6 walks.
Change in NYHA function class | baseline to 12 weeks
  changes in NYHA functional class.
Change in Right heart failure Severity | Baseline to 12 weeks
  Worsening right HF- defined as need for increase in diuretic dose or open-label initiation of a potassium sparing diuretic, or hospitalization or need for IV diuretics
Clinical Outcomes | 12 weeks
  Hospitalization and/or all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mielniczuk, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with researchers outside of Dr. Mielniczuk's research team.